CLINICAL TRIAL: NCT02368977
Title: Third Eye Panoramic Device Feasibility Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Avantis Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Avantis TEP 13-01
Record Dates: First submitted 2015-02-11; First posted 2015-02-23 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
Keywords: Colonoscopy; Polyps; Adenomas
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Adenoma

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will undergo examination with a Third Eye Panoramic device in conjunction with a standard colonoscope to evaluate the feasibility of using the study device to provide video imaging of areas of the colon that are difficult to evaluate with the colonoscope alone.
  Interventions: Device: Third Eye Panoramic device

INTERVENTIONS:
Device: Third Eye Panoramic device — A Third Eye Panoramic device will be attached to the tip of the colonoscope and will provide two additional views from laterally-oriented video cameras during the colonoscopy procedure.

SUMMARY:
This study will evaluate the feasibility of using the Third Eye Panoramic device in conjunction with standard colonoscopes in a clinical setting.

Patients will undergo a colonoscopy procedure during which the study device will provide video imaging of areas of the colon that are difficult to evaluate with the colonoscope alone.

The utility of the device will be assessed from the impressions of the investigators and from telephone follow-up with subjects to assess for post-procedural complications.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility of using the Third Eye Panoramic device along with a standard colonoscope as a means of enhancing the ability of endoscopists to view areas that are hidden from the view of the colonoscope.

Colonoscopy is generally agreed to be the best method for detecting and removing cancers and pre-cancerous adenomas in the colon. However, numerous studies have demonstrated that from 22% to over 40% of adenomas are missed during standard colonoscopy. More importantly, 12% of large adenomas (at least 1 cm) are missed even by expert endoscopists using meticulous technique with the best available equipment, and these large adenomas are the ones that are most likely to transform into cancer.

Factors such as quality of bowel cleansing and time spent examining the colonic mucosa have been shown to affect miss rates. However, comparison with the results of CT colonography has shown that 2/3 of missed adenomas are located behind folds in the wall of the colon, in areas that are very difficult to see with a standard forward-viewing colonoscope.

When clipped onto the tip of a standard colonoscope, the Third Eye Panoramic device provides two additional miniature video cameras and light sources that offer views to the left side and right side of the colonoscope's tip. These lateral views complement the forward view of the colonoscope's camera to result in a "panoramic" view of over 300°. This extreme wide-angle view allows the endoscopist to examine the areas located behind folds.

In this study, each subject will undergo a colonoscopy procedure utilizing the Third Eye Panoramic device along with a standard colonoscope.

The investigators will evaluate issues related to usability and safety based on their experience and impressions, with telephone follow-up with subjects to assess for any post-procedural complications.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup.
2. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Patients >75 years of age;
2. Patients with a history of colonic resection;
3. Patients with suspected chronic stricture potentially precluding complete colonoscopy;
4. Patients with diverticulitis or toxic megacolon;
5. Patients with a history of radiation therapy to abdomen or pelvis;
6. Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11-12 (Actual); Primary Completion 2017-10-11 (Estimated); Study Completion 2017-10-11 (Estimated)

PRIMARY OUTCOMES:
Device usability factors | 1 hour (average duration of procedure)
  Device usability as measured by investigators' qualitative impressions regarding ease of use and any potential interference with function of colonoscope.

SECONDARY OUTCOMES:
Device video factors | 1 hour (average duration of procedure)
  Video image quality and ability to view areas behind folds as measured by investigators' qualitative impressions
Patient safety assessed by number of subjects with adverse events as a measure of safety and tolerability | At time of procedure and up to 48 hours after completion of procedure
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Rubin, MD, Principal Investigator — New York Hospital Queens - Weill Cornell Medical College
Locations (1):
- New York Hospital Queens, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rubin M, Lurie L, Bose K, Kim SH. Expanding the view of a standard colonoscope with the Third Eye Panoramic cap. World J Gastroenterol. 2015 Oct 7;21(37):10683-7. doi: 10.3748/wjg.v21.i37.10683. PMID 26457029